CLINICAL TRIAL: NCT00744016
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Use of Mesalamine Pellet Formulation 1.5G QD to Maintain Remission From Mild to Moderate Ulcerative Colitis
Brief Title: Mesalamine Pellet Formulation to Maintain Remission of Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Audrey Shaw, Ph.D, Salix Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MPUC3003
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Ulcerative Colitis
Keywords: UC; Ulcerative colitis; IBD; Inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 1 (Active Comparator): Granulated mesalamine
  Interventions: Drug: Granulated mesalamine

INTERVENTIONS:
Drug: Granulated mesalamine — 0.375 g of mesalamine granules were encapsulated in a hard gelatin shell. 1.5 g of eMG (4 capsules) were administered orally QD, in the morning
  Other Names: mesalamine pellets
  Arms: 1
Drug: Placebo — Matching placebo capsules (4 capsules) were administered orally QD, in the morning
  Arms: 2

SUMMARY:
The purpose of this study is to compare the maintenance of mild to moderate ulcerative colitis remission with six months of treatment with 1.5 grams of mesalamine pellets each day versus placebo.

DETAILED DESCRIPTION:
This is a phase 3, multicenter, double-blind, randomized, placebo controlled study evaluating the effectiveness and safety of eMG 1.5 g given once daily (QD) compared with placebo in approximately 300 subjects with demonstrated remission from UC. Eligible subjects are randomized in a 2:1 ratio (active:placebo) to receive 1 of 2 treatments: 1.5g eMG QD (four capsules total) or matching placebo capsules QD for 6 months.

The study consists of a Screening phase (completed within 7 days prior to randomization), a Treatment phase (6 months), and a Follow-up visit (2 weeks after end-of-study [EOS] visit). The Treatment phase consists of 4 scheduled study visits: Visit 1 (Baseline)/Randomization (Day 1), Visit 2 (Month 1), Visit 3 (Month 3), Visit 4/EOS (Month 6).

Primary objective:

To compare the maintenance of remission from mild to moderate ulcerative colitis (UC) as measured by rectal bleeding and endoscopic mucosal appearance after 6 months of treatment with encapsulated mesalamine granules (eMG) at 1.5 g QD, as compared with placebo.

Secondary objective:

To compare the safety and tolerability of long-term dosing with eMG at 1.5 g QD as compared with placebo in the maintenance of remission from mild to moderate UC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ulcerative colitis and in remission for at least 1 month.
* Greater than 18 years of age.

Exclusion Criteria:

* Allergy/intolerance to aspirin, mesalamine or other salicylates.
* Prior bowel surgery other than appendectomy.
* Pregnancy, at risk of pregnancy or lactating.
* HIV or hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who were relapse free after 6 months of treatment. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Audrey L Shaw, Ph.D., Study Director — Bausch Health Americas, Inc.
Locations (1):
- Bristol, Connecticut, United States

REFERENCES:
- [Derived] Zakko SF, Gordon GL, Murthy U, Sedghi S, Pruitt R, Barrett AC, Bortey E, Paterson C, Forbes WP, Lichtenstein GR. Once-daily mesalamine granules for maintaining remission of ulcerative colitis: pooled analysis of efficacy, safety, and prognostic factors. Postgrad Med. 2016;128(3):273-81. doi: 10.1080/00325481.2016.1152876. Epub 2016 Mar 1. PMID 26861051
- [Derived] Lichtenstein GR, Gordon GL, Zakko S, Murthy U, Sedghi S, Pruitt R, Barrett AC, Bortey E, Paterson C, Forbes WP. Long-Term Benefit of Mesalamine Granules for Patients Who Achieved Corticosteroid-Induced Ulcerative Colitis Remission. Dig Dis Sci. 2016 Jan;61(1):221-9. doi: 10.1007/s10620-015-3866-7. Epub 2015 Nov 12. PMID 26563167
- [Derived] Lichtenstein GR, Zakko S, Gordon GL, Murthy U, Sedghi S, Pruitt R, Merchant K, Bortey E, Forbes WP. Mesalazine granules 1.5 g once-daily maintain remission in patients with ulcerative colitis who switch from other 5-ASA formulations: a pooled analysis from two randomised controlled trials. Aliment Pharmacol Ther. 2012 Jul;36(2):126-34. doi: 10.1111/j.1365-2036.2012.05142.x. Epub 2012 May 23. PMID 22617015